CLINICAL TRIAL: NCT01303146
Title: and Safety of METAZYM (Recombinant Human Arylsulfatase A or rhASA) for the Treatment of Patients With Late Infantile MLD Who Had Previously Hematopoietic Stem Cell Transplantation
Brief Title: Efficacy METAZYM for the Treatment Metachromatic Leukodystrophy Treated With Hematopoietic Stem Cell Transplantation
Acronym: Azylis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: European Leukodystrophy Association (Other); Zymenex A/S (Industry); Shire (Industry)
Responsible Party: VACHER Yannick, Department of Clinical Research of developpement
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P070805
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Metachromatic Leukodystrophy
Keywords: Metachromatic Leukodystrophy; Enzyme replacement therapy; Allogeneic hematopoietic stem cell transplantation
MeSH Terms: conditions — Leukodystrophy, Metachromatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enzyme replacement therapy (Experimental): intravenous infusion 100U/kg every other week for 18 months
  Interventions: Drug: rhARSA

INTERVENTIONS:
Drug: rhARSA — intravenous infusion 100U/kg every other week for 18 months
  Other Names: HGT-1111; Metazym

SUMMARY:
There is currently no effective treatment for late infantile MLD once clinical symptoms are evident. METAZYM is a recombinant human arylsulfatase A developed for an intravenous ERT for the treatment of late infantile MLD. The overall objective of this study is to evaluate the efficacy and safety of intravenous rhASA treatment in a patient with late infantile MLD who had previously received hematopoietic stem cell transplantation (HCT).

DETAILED DESCRIPTION:
Metachromatic Leukodystrophy (MLD) is a rare autosomal recessive disorder caused by the deficiency of the Arylsulfatase A enzyme (ARSA), resulting in accumulation of galactosyl sulfatide (cerebroside sulfate), a major constituent of the myelin sheath. Accumulation of galactosyl sulfatides leads to a progressive degeneration of the white matter in the central and peripheral nervous system (CNS, PNS) and neuronal degeneration. The late infantile form of MLD, which usually is diagnosed in the second year of life, is the most frequent and severe form of the disease. The prognosis is severe, leading to vegetative stage or death within few years after the diagnosis. There is no treatment for patients affected with this early onset form of the disease. In patients with late-onset MLD (juvenile and adult forms), allogeneic hematopoietic stem cell transplantation can stabilize the cerebral demyelination. This treatment is however inefficient in patients with late infantile MLD at a symptomatic stage. The overall objective is to evaluate the efficacy and safety of rhASA treatment in a patient with late infantile MLD who had received HCT at a presymptomatic stage of the disease. Patient will receive rhARSA (100 U/kg) intravenously every other week for a period of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject's legally authorized guardian(s) must provide signed, informed consent prior to performing any study-related activities.
* The patient must have a confirmed diagnosis of MLD as defined by:ARSA activity < 10 nmol/h/mg in leukocytes prior to HCT; Presence of elevated sulfatide in urine prior to HCT
* The patient must have a residual level of voluntary function (as judged by the investigator), including presence of residual cognitive function (attention, executive and visual functions) as well as the presence of residual voluntary motor function in one upper or lower limb as a minimum.
* The patient must have an age at the time of screening ≥ 6 months
* The patient must have had onset of symptoms before the age of 4 years
* The subject and his/her guardian(s) must have the ability to comply with the clinical protocol
* The patients' medical record must document that the legal guardian(s) has had independent counselling or a consultation regarding stem cell transplantation in order to assure that the guardian(s) is fully informed regarding the risks and benefits of this alternative

Exclusion Criteria:

Patient will be excluded from this study if they do not meet the specific inclusion criteria, or if any of the following criteria apply:

* Presence of a gross motor function measure (GMFM < 25)
* Presence of severe pseudo-bulbar signs (weakness and disco-ordination of tongue and swallowing muscles leading to severe difficulty with swallowing)
* Spasticity so severe to inhibit transportation
* Known multiple sulfatase deficiency
* Presence of major congenital abnormality
* Presence of known chromosomal abnormality and syndromes affecting psychomotor development
* Presence of known clinically significant cardiovascular, hepatic, pulmonary or renal disease or other medical condition
* Any other medical condition or serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, would preclude participation in the trial
* Use of any investigational product within 30 days prior to study enrolment or currently enrolled in another study which involves clinical investigations
* Received ERT with rhASA from any source

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of METAZYM on peripheral nerve function by electrophysiological studies (motor and sensory nerves conduction velocities) every 6 months; | every 6 months
Efficacy of METAZYM on peripheral nerve sulfatide storage and demyelination by nerve biopsy at baseline and week 26; | week 26
Efficacy of METAZYM on functional capacity by assessing motor function (GMFM) every 6 months | every 6 months

SECONDARY OUTCOMES:
Efficacy of METAZYM on central nervous system involvement by evaluation of cognitive and neurological function, somatosensory and auditory evoked potentials, and brain MRI every 6 months; | every 6 months
Safety profile of METAZYM by monitoring AE's, vital sign parameters and physical examination findings before each injection, as well as ECGs and routine clinical laboratory tests every 3 months. | every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Aubourg, MD, PhD, Study Chair — Department of Pediatric Endocrinology and Neurology, Saint Vincent de Paul Hospital, Paris
Locations (1):
- Department of Pediatric Endocrinology and Neurology, Saint Vincent de Paul Hospital, Paris, France